CLINICAL TRIAL: NCT04993066
Title: Clinical Evaluation to Assess the Safety and Efficacy of GentleMax Pro/ GentleMax Pro Plus
Brief Title: Clinical Evaluation to Assess the Safety and Efficacy of GentleMax Pro Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMP19002, phase II
Record Dates: First submitted 2021-07-19; First posted 2021-08-06 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Pseudofolliculitis Barbae; Unwanted Hair; Pigmented Lesions; Vascular Lesion; Onychomycosis; Wrinkle; Acne
MeSH Terms: conditions — pseudofolliculitis barbae; Onychomycosis; Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Arm (Experimental): All study subjects are to receive treatment with GentleMax Pro Plus device. Subjects will be scheduled to receive as little as one (1) and up to eight (8) treatments with the GentleMax Pro Plus™ Laser System. Up to 2 follow-ups will occur.
  Interventions: Device: GentleMax Pro Plus

INTERVENTIONS:
Device: GentleMax Pro Plus — The GentleMax Pro Plus laser system to be used in this study received 510(k) market clearance from the U.S. Food and Drug Administration (FDA) under K201111 on May 26, 2020

SUMMARY:
Demonstrate the safety and efficacy of the GentleMax Pro Plus™ laser system for its intended uses: hair removal including pseudofolliculitis barbae (PFB), clearance of pigmented and/or vascular lesions, temporary increase of clear nail in patients with onychomycosis and improvement in appearance of wrinkles. Evaluate GentleMax Pro Plus™ laser system for the clearance of acne.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older
2. Willingness to provide signed, informed consent to participate in the study
3. Presence of unwanted hair, moderate or greater benign pigmented lesions, active acne, vascular lesions, nails affected with onychomycosis, and/or wrinkles assessed as Fitzpatrick Wrinkle and Elastosis Score (FWS) >/= 1
4. Willingness to adhere to study treatment and follow-up schedule
5. Willingness to adhere to post-treatment care instructions
6. Willingness to allow photographs and/or video of treated areas, and to release their use for scientific/educational and/or promotional/marketing purposes
7. Willing to abstain from any other procedures, medications or topicals in the study treatment areas for the duration of the study which the investigator deems would interfere with the study

Exclusion Criteria:

1. Pregnant, planning pregnancy during the study, or breast feeding
2. Blonde, grey, or white hair in subjects seeking hair removal
3. Tattooed skin in the intended treatment area
4. Active sun tan in the intended treatment area
5. History of active Herpes Virus Simplex (HSV) or similar condition in the intended treatment area unless treated with prophylactic medication
6. History of melanoma
7. History of vitiligo in the intended treatment area
8. History of keloid or hypertrophic scar formation
9. History of Melasma in the intended treatment area or per Investigator's discretion
10. Severe immunosuppression resulting from medications and/or a medical condition that could impair healing after treatment
11. Open wound or infection in the intended treatment area
12. History of light induced seizure disorders
13. The subject is not suitable, in the opinion of the Investigator, for participation in the study due to inability to adhere to the study requirements, medical, or other reasons that could compromise the study integrity or subject safety
14. Dermatologic and/or cosmetic procedures including use of medications, or topicals in the intended treatment area(s) during a timepoint prior to the study that the investigator deems the subject unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Treatment Time | 8 Months
  Evaluate the speed (time of treatment completion) with larger spot sizes for hair removal
Hair Count Assessments | 14 Months
  Improvement in hair clearance quantified by hair counts taken within a portion of the treatment area and percent reduction by assessments of digital photos taken at Baseline compared to follow-ups.
Global Aesthetic Improvement Score | 7 Months
  Improvement in the appearance of wrinkles, benign pigmented lesions, and/or vascular lesions from baseline to follow-up(s) via the Investigator Global Aesthetic Improvement Score (IGAIS) whereas 1 = very much improved and 5 = worse. A lower score post treatment(s) indicates a better outcome.
Fitzpatrick Wrinkle and Elastosis Score | 7 Months
  Improvement in the appearance of wrinkles from baseline to follow-up(s) via the Investigator Fitzpatrick Wrinkle and Elastosis Scale whereas 1 = fine wrinkles and mild elastosis and 9 = deep wrinkles and severe elastosis. A lower score post treatment(s) indicates a better outcome.
Pigment Improvement Score | 7 Months
  Improvement in BPLs from baseline to follow-ups via the Investigator Pigment Improvement Score (PIS) whereas 0 = no improvement and 4 = excellent response. A higher score post treatment(s) indicates a better outcome.
Acne Counts | 5 Months
  Measured by improvement of acne counts from baseline compared to follow-ups. A lower score post treatment(s) indicates a better outcome.
Onychomycosis Score | 9 Months
  Improvement in the appearance of nails from Baseline to follow-up(s) via the Scoring Clinical Index of Onychomycosis (SCIO Index) which ranges from 0 to 30 whereas 0 indicates lesser degree of onychomycosis and 30 indicates higher degree of onychomycosis. A lower score post treatment(s) indicates a better outcome.
Onychomycosis Score | 9 Months
  Improvement in the appearance of nails from Baseline to follow-up(s) via the Onychomycosis Improvement Scale whereas 1 = completely cleared and 5 = worse. A lower score post treatment(s) indicates a better outcome.

SECONDARY OUTCOMES:
Subject Satisfaction Score | 24 Months
  Overall subject satisfaction with study treatments per treatment indication as measured by Subject Satisfaction Scale whereas 1 = not satisfied and 5 = very satisfied. A higher score post treatment(s) indicates a better outcome.
Subject Global Aesthetic Improvement Score | 24 Months
  Overall subject improvement with study treatments per treatment indication as measured by Subject Global Aesthetic Improvement Score (SGAIS) whereas 1 = very much improved and 5 = worse. A lower score post treatment(s) indicates a better outcome.
Subject Pain | 8 Months
  Measurement of Subject Pain Assessment post-treatment for all subjects, using an 11-point pain Numerical Rating Scale where 0=no pain, 10=extreme pain

CONTACTS AND LOCATIONS:
Locations (1):
- Candela Institute of Excellence, Marlborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
N/A, no plan to share IPD